CLINICAL TRIAL: NCT04122547
Title: Efficacy of Roflumilast on Exacerbations in Patients With Non-cystic Fibrosis Bronchiectasis: a Randomized Double-blind Placebo-controlled Trial
Brief Title: Efficacy of Roflumilast on Exacerbations in Patients With Non-cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Siwasak Juthong, Clinical Professor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25132558
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Exacerbation Copd; Bronchiectasis; Lung Function Decreased
Keywords: Bronchiectasis; roflumilast; exacerbation; lung function
MeSH Terms: conditions — Bronchiectasis; Respiratory Insufficiency | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Roflumilast (Active Comparator): Roflumilast 500 microgram one tab oral per day
  Interventions: Drug: Roflumilast
- Placebo (Placebo Comparator): One tablet oral per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — Active drug
  Other Names: Daxas
  Arms: Roflumilast
Drug: Placebo — Placebo one tablet oral od
  Arms: Placebo

SUMMARY:
Roflumilast compare with placebo for decrease infected exacerbation in non-cystic Bronchiectasis

DETAILED DESCRIPTION:
Efficacy and RCT compare roflumilast vs placebo for 6 months in frequent infectious exacerbation in non-cystic bronchiectasis in Thailand

ELIGIBILITY:
Inclusion Criteria:

* symptomatic Bronchiectasis
* history at least 2 exacerbation last year

Exclusion Criteria:

* comorbidity with chronic obstructive pulmonary disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
acute deterioration of of bronchiectasis symptoms | 6 months
  acute dyspnea worsening respiratory of symptoms

SECONDARY OUTCOMES:
Lung functions | 6 months
  FEV1
Exercise capacity | 6 months
  6 minute walk distance

OTHER OUTCOMES:
Health related Quality of life | 6 months
  SGRQ scores, score range from 0-80, high score mean more symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Kanung Saejiam, MS, Study Director — Prince of Songkla University
Locations (1):
- Songklanagarind hospital, Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No